CLINICAL TRIAL: NCT07253428
Title: IMPACT OF SUGAMADEX ON AGITATION UPON EMERGENCE FOLLOWING ADULT NASAL SURGERIES.
Brief Title: Emergence Agitation
Acronym: Sugamadex
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sabah Nageeb, Lecturer of anesthesia and intensive care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KASC-KSA; SABAHNAGEEB (Other: KING SALMAN SPECIALIST HOSPITAL)
Record Dates: First submitted 2025-11-16; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Emergence Agitation; Nasal Surgery
Keywords: Sugamadex,; Neostigmine; anesthesia recovery; nasal surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Neostigmine; Atropine

STUDY DESIGN:
Intervention Model Description: Sugamadex group will receive sugamadex as a reversal agent of the muscle relaxant; rocuronium. the aim is to study the impact of adequate muscle relaxation upon the emergence agitation. This will be compared the neostigmine group which will receive it as a reversal agent of the muscle relaxation
Masking Description: no need for masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugamadex group (Active Comparator): Sugamadex group will receive sugamadex as a reversal agent of the muscle relaxant; rocuronium
  Interventions: Drug: Sugamadex
- Neostigmine group (Other): Neostigmine group will receive the neostigmine as a reversal of the muscle relaxant; rocuronium
  Interventions: Drug: Neostigmine + Atropine

INTERVENTIONS:
Drug: Neostigmine + Atropine — Neostigmine group will receive the neostigmine as a reversal of the muscle relaxant; rocuronium
  Other Names: N.group
  Arms: Neostigmine group
Drug: Sugamadex — Sugamadex group will receive sugamadex as a reversal agent of the muscle relaxant; rocuronium Neostigmine group will receive the neostigmine as a reversal of the muscle relaxant; rocuronium.
  Both interventions will be used to compare the effect of adequate muscle relaxation upon the emergence agitation.
  Other Names: S.group
  Arms: Sugamadex group

SUMMARY:
The impact of sugammadex on agitation upon emergence following adult nasal surgeries is an issue which needs to be studied that links anesthetic management with postoperative recovery.

DETAILED DESCRIPTION:
The included patients in the study will not be premedicated by sedatives, they will be preoxygenated for 5 minutes by 100% oxygen. The induction of anesthesia will be by fentanyl 100 microgram, 1.5 mg/kg lidocaine followed by propofol 2mg/kg, and rocuronium 0.5 mg/kg. oral intubation will be commenced and an oral pack will be inserted. Anesthesia will be maintained by sevoflurane 2% and N2O : O2 ratio of 50: 50.

Hypotensive anesthesia will be conducted by labetalol 10- 20 mg i.v. At the end of surgery inhalational anesthesia will be abandoned and muscle relaxant will be antagonized either by sugamadex 1mg/kg or neostigmine 0.05 mg/kg mixed with atropine 0.02 mg/kg. After awakening of the of the patients, emergence agitation will be assessed by Agitation and Emergence Score (AES): This scale is ranging from 0 (calm and cooperative) to 4 (combative, aggressive behavior).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aging from 18 to 60 years old, undergoing nasal surgeries such as septoplasty, FESS or Rhinoplasty
* ASA I and ASA II

Exclusion Criteria:

* Patients receiving any medications which may affect recovery state e.g. Antipsychotics.
* Smokers
* Obstructive sleep apnea patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 486 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of emergence agitation following adult nasal surgeries in patients receiving sugammadex versus a traditional neuromuscular blocking agent reversal method. | perioperative
  Agitation and Emergence Score (AES): This scale is ranging from 0 (calm and cooperative) to 4 (combative, aggressive behavior).

SECONDARY OUTCOMES:
duration to full consciousness | Perioperative
  Minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Rabah Alharbi, Hail, Saudi Arabia